CLINICAL TRIAL: NCT01084174
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study of Sublingual/Oral Immunotherapy for the Treatment of Peanut Allergy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00032256
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Peanut Hypersensitivity; Food Hypersensitivity; Immediate Hypersensitivity
Keywords: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity; Hypersensitivity, Immediate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active SLIT/Placebo OIT (Experimental): These subjects will receive peanut powder given orally and placebo extract given sublingually.
  Interventions: Drug: Peanut powder; Drug: Placebo extract
- Active OIT/Placebo SLIT (Experimental): These subjects will receive peanut extract given sublingually and placebo powder given orally.
  Interventions: Drug: Peanut extract; Drug: Placebo powder

INTERVENTIONS:
Drug: Peanut powder — Delivered orally
  Arms: Active SLIT/Placebo OIT
Drug: Peanut extract — Delivered sublingually
  Arms: Active OIT/Placebo SLIT
Drug: Placebo extract — Delivered sublingually
  Arms: Active SLIT/Placebo OIT
Drug: Placebo powder — Delivered orally
  Arms: Active OIT/Placebo SLIT

SUMMARY:
The purpose of this study is to explore the safety and efficacy of a sublingual (under the tongue) immunotherapy (SLIT) dosing regimen and an oral immunotherapy (OIT) regimen in inducing desensitization and long term tolerance in children with persistent peanut allergy.

DETAILED DESCRIPTION:
To effectively address the Primary Objectives of this pilot study, 30 subjects aged 6-21 years with: (1) a convincing clinical history of peanut allergy (PA), (2) a serum immunoglobulin E (IgE) specific to peanut of >0.35 kilo units per liter (kU/L) and a skin prick test (SPT) wheal >3 mm, will be enrolled. Subjects will be recruited from the Johns Hopkins Pediatric Allergy Clinic.

Participants will undergo an initial screening visit that will include a medical history, physical exam, skin testing, and phlebotomy. Informed consent and assent will be obtained. At the next two visits, 20 participants will complete a double-blind placebo-controlled food challenge (DBPCFC). Eligible subjects will be randomized in a 1:1 ratio into two groups. One group will receive active SLIT with placebo OIT and the other group will begin active OIT with placebo SLIT dose escalation. Over the next 16 weeks of the study, subjects will undergo SLIT and OIT dose increases. A maintenance dose will then be taken at home daily for 12 months. A DBPCFC will be completed after 6 months and 12 months of home dosing. Those patients who pass the DBPCFC will be taken off SLIT and OIT for 4 weeks. A final challenge will be administered at the end of this period.

Ten additional peanut-allergic subjects age 6-21 years will be enrolled and followed as longitudinal controls for the mechanistic studies. These subjects will follow a modified schedule compared to those subjects receiving study treatment and will be evaluated by phlebotomy, end point titration prick skin testing, and saliva collection. These patients will continue strict avoidance of peanut unless otherwise advised by their personal physician.

ELIGIBILITY:
Inclusion Criteria:

* Are ages 6 to 21 years of either sex, any race, and any ethnicity at the time of the initial visit.
* Have a physician diagnosed peanut allergy or a convincing clinical history of peanut allergy (urticaria, upper or lower respiratory symptoms, GI disturbances, rash or oral symptoms).
* Have a skin prick test positive to peanut (diameter of wheal 3 mm ≥ negative control) and detectable serum peanut-specific IgE level (UniCAP ≥ 0.35 kU/L).
* Have a positive reaction to a cumulative dose of ≤1,000 mg of peanut powder in the initial qualifying DBPCFC.
* Use an effective method of contraception by females of childbearing potential to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of their participation in the study.
* Ability to perform spirometry maneuvers in accordance with the American Thoracic Society (ATS) guidelines (1994).
* Have self-injectable epinephrine (i.e. EpiPen® or EpiPen Jr.®) available at all times.
* Provide signed informed consent (by parent or legal guardian if the subject is a minor) and informed assent if applicable.

Exclusion Criteria:

* Have a history of severe anaphylaxis to peanut with hypoxia (cyanosis or peripheral capillary oxygen saturation (SpO2) ≤92% at any stage), hypotension or neurological compromise (confusion, collapse, loss of consciousness or incontinence).
* Tolerates more than 1,000 mg of peanut powder at the initial qualifying DBPCFC.
* Have a viral upper respiratory infection (URI) or gastroenteritis within 7 days of OFC (OFC will need to be rescheduled).
* Currently participating in a study using an investigational new drug.
* Participation in any interventional study for the treatment of food allergy in the past 12 months.
* Pregnancy or lactation
* Allergy to placebo ingredients (Glycerin or oat flour) OR reacts to any dose of placebo during the qualifying OFC.
* Currently in a buildup phase of any allergy immunotherapy.
* Poor control of atopic dermatitis.
* Have pulmonary function tests with forced expiratory volume 1 (FEV1) value <80% predicted or any clinical features of greater than moderate persistent asthma and greater than high daily doses of inhaled corticosteroids (>500µg/day fluticasone or equivalent).
* Use of steroid medications (oral steroids, such as prednisone or Medrol, steroid injections, such as Kenalog, or IV or oral corticosteroid burst) in the following manners:

  o History of daily oral steroid dosing within 4 weeks prior to baseline visit or for > 1 month during the past year or burst oral steroid course in the past 6 months or > 1 burst oral steroid course in the past year.
* Asthma requiring

  * ≥1 hospitalization in the past year for asthma or
  * >1 ER visit in the past 6 months for asthma
* Use of omalizumab or other non-traditional forms of allergen immunotherapy (e.g., oral or sublingual) or immuno-modulatory therapy (not including corticosteroids) or biologic therapy within the past year.
* Use of β-blockers (oral), angiotensin-converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARB), calcium channel blockers or tricyclic antidepressant therapy.
* Inability to discontinue antihistamines for 5 days for long acting and 3 days for short acting prior to skin testing or OFC's.
* History of alcohol or drug abuse.
* Active eosinophilic gastrointestinal disease in the past two years.
* Have other significant medical conditions (e.g., liver, gastrointestinal, kidney, cardiovascular, pulmonary disease, or blood disorders) which, in the opinion of the Investigator, make the subject unsuitable for induction of food reactions.
* Any previous intubation due to allergies or asthma.
* Severe reaction at initial DBPCFC, defined as:

  * Life-threatening anaphylaxis
  * Requiring overnight hospitalization

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2010-03; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Narisety SD, Frischmeyer-Guerrerio PA, Keet CA, Gorelik M, Schroeder J, Hamilton RG, Wood RA. A randomized, double-blind, placebo-controlled pilot study of sublingual versus oral immunotherapy for the treatment of peanut allergy. J Allergy Clin Immunol. 2015 May;135(5):1275-82.e1-6. doi: 10.1016/j.jaci.2014.11.005. Epub 2014 Dec 18. PMID 25528358

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active SLIT/Placebo OIT | Active OIT/Placebo SLIT
Started | 10 | 11
Completed | 9 | 7
Not Completed | 1 | 4
Not completed — gastrointestinal symptoms | 1 | 1
Not completed — Eosinophilic esophagitis | 0 | 1
Not completed — Anaphylaxis | 0 | 1
Not completed — Participant noncompliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active SLIT/Placebo OIT | Active OIT/Placebo SLIT | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 11 | 21
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21
Prior history of peanut anaphylaxis [Count of Participants; unit: Participants] | 1 | 6 | 7
Other food allergies [Count of Participants; unit: Participants] | 10 | 10 | 20
Atopic dermatitis [Count of Participants; unit: Participants] | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Induced Peanut Desensitization at 12 Months
Description: Peanut desensitization was defined as a greater than 10-fold increase in oral food challenge (OFC) threshold after 12 months of therapy.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active SLIT/Placebo OIT | Active OIT/Placebo SLIT
Number analyzed (Participants) | 9 | 7
Participants | 9 | 7

2. Secondary Outcome: Between Arm Change in IgG4 From Baseline to End of Dose Build-up (up to 16 Weeks)
Description: Serum immunoglobulin G4 (IgG4) levels are measured in milligrams of Antibody per liter (mga/L) and were collected at baseline and at the end of dose build-up (up to 16 weeks)
Time Frame: Baseline and end of dose build-up (up to 16 weeks)
Measure: Median (Full Range); unit: mga/L
Arm/Group | Active SLIT/Placebo OIT | Active OIT/Placebo SLIT
Number analyzed (Participants) | 10 | 11
mga/L
  Baseline | 0.9 [0.19 to 1.76] | 1.3 [0.22 to 5.89]
  End of dose build-up (up to 16 weeks) | 2.5 [0.47 to 7.07] | 11.3 [0.99 to 58.7]
Statistical Analysis 1: Comparison: Active SLIT/Placebo OIT vs Active OIT/Placebo SLIT; Test type: Other; p = .003, Regression, Linear; Analyzed by linear regression models using generalized estimating equations to account for repeated measures over time with robust standard errors

3. Secondary Outcome: Between Arm Change in IgG4 From Baseline to 6 Months
Description: IgG4 levels are measured in milligrams of Antibody per liter (mga/L) and were collected at baseline and at 6 months
Time Frame: Baseline and 6 months
Population: One participant in the Active sublingual immunotherapy (SLIT)/Placebo oral immunotherapy (OIT) arm and 4 participants in the Active OIT/Placebo SLIT arm discontinued prior to month 6.
Measure: Median (Full Range); unit: mga/L
Arm/Group | Active SLIT/Placebo OIT | Active OIT/Placebo SLIT
Number analyzed (Participants) | 9 | 7
mga/L
  Baseline | 0.9 [0.19 to 1.76] | 1.3 [0.22 to 5.89]
  6 months | 7.9 [1.51 to 76.2] | 83.4 [21.2 to 677]
Statistical Analysis 1: Comparison: Active SLIT/Placebo OIT vs Active OIT/Placebo SLIT; Test type: Other; p < .001, Regression, Linear

4. Secondary Outcome: Between Arm Change in IgG4 From Baseline to 12 Months
Description: IgG4 levels are measured in milligrams of Antibody per liter (mga/L) and were collected at baseline and at 12 months
Time Frame: Baseline and 12 months
Population: One participant in the Active SLIT/Placebo OIT arm and 4 participants in the Active OIT/Placebo SLIT arm discontinued prior to month 12.
Measure: Median (Full Range); unit: mga/L
Arm/Group | Active SLIT/Placebo OIT | Active OIT/Placebo SLIT
Number analyzed (Participants) | 9 | 7
mga/L
  Baseline | 0.9 [0.19 to 1.76] | 1.3 [0.22 to 5.89]
  12 months | 8.5 [2.42 to 69.1] | 76 [28.8 to 1790]
Statistical Analysis 1: Comparison: Active SLIT/Placebo OIT vs Active OIT/Placebo SLIT; Test type: Other; p < .001, Regression, Linear

5. Secondary Outcome: Between Arm Change in IgE From Baseline to End of Dose Build-up (up to 16 Weeks)
Time Frame: Baseline to end of dose build-up (up to 16 weeks)
Measure: Mean (Full Range); unit: kUa/L
Arm/Group | Active SLIT/Placebo OIT | Active OIT/Placebo SLIT
Number analyzed (Participants) | 9 | 7
kUa/L
  Baseline | 163 [37.5 to 746] | 169 [35.1 to 716]
  End of dose build-up (up to 16 weeks) | 369 [47.4 to 1960] | 392 [84 to 1069]
Statistical Analysis 1: Comparison: Active SLIT/Placebo OIT vs Active OIT/Placebo SLIT; Test type: Other; p = 0.40, Regression, Linear

6. Secondary Outcome: Between Arm Change in IgE From Baseline to 6 Months
Description: Serum immunoglobulin E (IgE) levels are measured in kilo units of Antibody per liter (kUa/L) and were collected at baseline and at 6 months
Time Frame: Baseline and 6 months
Measure: Median (Full Range); unit: kUa/L
Arm/Group | Active SLIT/Placebo OIT | Active OIT/Placebo SLIT
Number analyzed (Participants) | 9 | 7
kUa/L
  Baseline | 163 [37.5 to 746] | 169 [35.1 to 716]
  6 months | 387 [34.1 to 1032] | 68 [50.9 to 204]
Statistical Analysis 1: Comparison: Active SLIT/Placebo OIT vs Active OIT/Placebo SLIT; Test type: Other; p = .07, Regression, Linear

7. Secondary Outcome: Between Arm Change in IgE From Baseline to 12 Months
Description: IgE levels are measured in kilo units of Antibody per liter (kUa/L) and were collected at baseline and at 12 months
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: kUa/L
Arm/Group | Active SLIT/Placebo OIT | Active OIT/Placebo SLIT
Number analyzed (Participants) | 9 | 7
kUa/L
  Baseline | 163 [37.5 to 746] | 169 [35.1 to 716]
  12 months | 273 [21.0 to 1111] | 53 [32.4 to 82.9]
Statistical Analysis 1: Comparison: Active SLIT/Placebo OIT vs Active OIT/Placebo SLIT; Test type: Other; p = .007, Regression, Linear

ADVERSE EVENTS:
Groups:
- Active SLIT/Placebo OIT: Adverse event information is based on percentages of doses. There were 4578 total doses in the Active SLIT/Placebo OIT treatment arm
- Active OIT/Placebo SLIT: Adverse event information is based on percentages of doses. There were 4049 total doses in the Active OIT/Placebo SLIT treatment arm
Arm/Group | Active SLIT/Placebo OIT | Active OIT/Placebo SLIT
All-Cause Mortality (participants affected / at risk) | 0/4578 | 0/4049
Serious Adverse Events (participants affected / at risk) | 0/4578 | 0/4049
Other Adverse Events (participants affected / at risk) | 416/4578 | 1736/4049
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active SLIT/Placebo OIT (N=4578) | Active OIT/Placebo SLIT (N=4049)
Gastrointestinal symptoms (Gastrointestinal disorders) | 325 (325) | 1344 (1344) — including oral/pharyngeal symptoms
skin symptoms (Skin and subcutaneous tissue disorders) | 64 (64) | 113 (113)
Respiratory Symptoms (Respiratory, thoracic and mediastinal disorders) | 27 (27) | 279 (279)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No